CLINICAL TRIAL: NCT04778969
Title: Coronary Artery Disease Patients Treated With Percutaneous Coronary Intervention: Analysis of the Korean Nationwide Health Insurance Database
Brief Title: Kor PCI - CAD Patients Treated With PCI: Analysis of the Korean Nationwide Health Insurance Database
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Mo Yang, Professor, Seoul National University Hospital
Other Study IDs: E-2009-016-1154
Record Dates: First submitted 2021-01-13; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Drug-eluting Stents; Drug-coated Balloon
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: drug-eluting stent — A group of percutaneous coronary intervention (PCI) using drug-eluting stents (DES)
  Other Names: DES group
Device: drug-coated balloon — A group of percutaneous coronary intervention (PCI) using drug-coated balloon (DCB)
  Other Names: DCB group

SUMMARY:
Current Status and Prognosis of Coronary artery disease patients treated with coronary intervention - Analysis of the Korean Nationwide Health Insurance Database

DETAILED DESCRIPTION:
This is a retrospective study and is conducted for all patients who received percutaneous coronary intervention among cohorts registered with the National Health Insurance Service.

Primary outcome is all cause of mortality. Secondary outcomes are cardiovascular death, ischemic stroke, cerebral hemorrhage, admission due to gastrointestinal bleeding, and admission due to major bleedings.

ELIGIBILITY:
Inclusion Criteria:

* All coronary artery disease patients wih Korean NHIS (National Health Insurance Service)-listed PCI

Exclusion Criteria:

* non-specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All coronary artery disease patients wih Korean NHIS (National Health Insurance Service)-listed PCI Patients are selected based on the registered treatment insurance code.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
All cause of death | 10 years
  'All cause of death' will be recorded as number of participants with 'All cause of death'

SECONDARY OUTCOMES:
Cardiovascular death | 10 years
  'Cardiovascular death' will be recorded as number of participants with 'Cardiovascular death'
ischemic stroke | 10 years
  'ischemic stroke' will be recorded as number of participants with 'ischemic stroke'
Cerebral hemorrhage | 10 years
  'Cerebral hemorrhage' will be recorded as number of participants with 'Cerebral hemorrhage'
Admission due to gastrointestinal bleeding | 10 years
  'Admission due to gastrointestinal bleeding' will be recorded as number of participants with 'Admission due to gastrointestinal bleeding'
Admission due to major bleeding | 10 years
  'Admission due to major bleeding' will be recorded as number of participants with 'Admission due to major bleeding' Thismeasure is a composite outcome, which includes cerebral hemorrhage, admission due to gastrointestinal bleeding.

IPD SHARING:
Plan to Share IPD: No
Since this research is conducted with a national public institution, data cannot be shared.